CLINICAL TRIAL: NCT04113681
Title: Pilot Study: Geniculate Artery Embolization in Knee Osteoarthrosis.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Cengarle-Samak, Interventional radiologist, Maisonneuve-Rosemont Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Geniculate embolization.
Record Dates: First submitted 2019-10-01; First posted 2019-10-03 (Actual); Last update posted 2021-03-08 (Actual); Status verified 2021-03

CONDITIONS: Osteoarthritis, Knee
Keywords: Embolization, Osteoarthritis, Knee, Geniculate Artery
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Intervention Model Description: Patients will be stratified into two groups:
  * Group 1: Patients between 18-50 years old with KL grade 3-4
  * Group 2: Patients age 50 years old and over with KL grade 1-4
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Geniculate Artery Embolization Arm (Experimental): Single-arm prospective study of geniculate artery embolization for symptomatic knee osteoarthritis
  Interventions: Procedure: Geniculate Artery Embolization

INTERVENTIONS:
Procedure: Geniculate Artery Embolization — 1. Conscious sedation : midazolam and fentanyl
  2. Local anesthesia : Lidocaine 2% subcutaneous
  3. Retrograde or anterograde common femoral artery access - 4Fr introducer
  4. Sub-therapeutic anticoagulation (heparin 2000 IU IA)
  5. Lower extremity arteriography
  6. Selective and supra-selective catheterization of geniculate arteries supplying painful region of the knee
  7. If abnormal arterial blushes are demonstrated selective and supra-selective embolization will be performed with Embozene microspheres (100 microns to 200 microns) - cold saline or ice-packs sac to be applied to overlying skin if significant cutaneous arteries are demonstrated at angiography.
  8. Angiographic end-points: embolization of abnormal blush while preserving the parent vessel
  9. Arteriotomy closure (manual compression or closure device)

SUMMARY:
Geniculate Artery Embolization (GAE) has recently been described and studied as a palliative treatment for osteoarthrosis-related knee pain in patients un-eligible for surgical intervention. This treatment is based on the hypothesis that hypervascularization and associated increased nerve proliferation are possible sources of chronic pain following the morphological changes of osteoarthrosis. A large animal model has shown digital subtraction arteriography to be well correlated to both the histological findings of synovial inflammation and synovial contrast enhancement on magnetic resonance imaging. This embolization technique has also been applied to other regions of the musculoskeletal system including the elbow and the shoulder.

DETAILED DESCRIPTION:
Primary Objective Confirm the efficacy and the effectiveness of geniculate artery embolization for pain control in knee osteoarthrosis.

Secondary Objective Evaluate the effectiveness of geniculate artery embolization for pain control in specific population: young patients between 18 and 50 years old with advanced osteoarthritis (KL grade 3 or 4) for whom an orthopedic surgeon has deemed a total knee arthroplasty is not an appropriate therapy, and whom have failed conservative management for at least 6 months.

Investigators propose a prospective pilot study on 40 patients with osteoarthrosis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years and older
* Moderate to severe knee pain (visual analog scale (VAS) > 70 mm)
* Pain refractory to at least 6 months of conservative therapies (anti-inflammatory drugs, or physical therapy, or muscle strengthening, or intra-articular injections)
* Localized pain on physical examination
* Kellgren-Lawrence (KL) Score on knee X-Ray
* Patients 50 years old and over : grade 1, 2, 3 or 4
* 18-50 years old: KL grade 3 or 4

Exclusion Criteria:

* Current local infection
* Life expectancy less than 6 months
* Known advanced atherosclerosis
* Rheumatoid or infectious arthritis
* Prior knee surgery
* Uncorrectable coagulopathy including international normalized ratio (INR) > 1.5 or platelets < 50,000
* Iodine allergy
* Renal dysfunction as defined by GFR < 60ml/min obtained within the past 30 days.
* Diabetic patient
* Previous embolization of the geniculate arteries during the last year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-14 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain control VAS | 12 months
  The pain intensity is assessed using VAS (horizontal line 100 mm in length). Subjects mark the VAS with a single vertical line to indicate their current pain level, with 0 mm representing "No Pain" and 100 mm representing "Worst Possible Pain".
  * Expected mean VAS pre treatment: 7
  * Expected mean VAS at 1, 3, 6 and 12 months: 3-4 (50% reduction)

SECONDARY OUTCOMES:
Function | 12 months
  Western Ontario and McMaster University Osteoarthritis Index (WOMAC) Subcategories of pain (5 items), stiffness (2 items), and physical function (17 items). Individuals select the level of difficulty they have performing various tasks using a 5 points Likert scale (0=None, 1=Slightly, 3=Very, 4=Extremely). Results are scored with a total maximum score of 96. A higher score indicates more difficulty in each of the categories.
  * Expected mean WOMAC score pre treatment: 50
  * Expected mean WOMAC score at 1, 3, 6 and 12 months: 25 (50% reduction).
Radiological examinations | 12 months
  * Knee x-ray examinations
  * Knee MRI (if a complication is suspected clinically)
  * Sustained response expected to be less likely with increased KL grade

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Cengarle-Samak, MD, Principal Investigator — CIUSSS de l'Est-de-l'Ile-de-Montreal
Locations (1):
- CIUSSS de l'Est-de-l'Île-de-Montréal, Installation Hopital Maisonneuve-Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] van Baardewijk LJ, Hoogeveen YL, van der Geest ICM, Schultze Kool LJ. Embolization of the Geniculate Arteries Is an Effective Treatment of Recurrent Hemarthrosis Following Total Knee Arthroplasty That Can Be Safely Repeated. J Arthroplasty. 2018 Apr;33(4):1177-1180.e1. doi: 10.1016/j.arth.2017.11.002. Epub 2017 Nov 24. PMID 29224993
- [Background] Bagla S, Rholl KS, van Breda A, Sterling KM, van Breda A. Geniculate artery embolization in the management of spontaneous recurrent hemarthrosis of the knee: case series. J Vasc Interv Radiol. 2013 Mar;24(3):439-42. doi: 10.1016/j.jvir.2012.11.011. PMID 23433418
- [Background] Okuno Y, Korchi AM, Shinjo T, Kato S, Kaneko T. Midterm Clinical Outcomes and MR Imaging Changes after Transcatheter Arterial Embolization as a Treatment for Mild to Moderate Radiographic Knee Osteoarthritis Resistant to Conservative Treatment. J Vasc Interv Radiol. 2017 Jul;28(7):995-1002. doi: 10.1016/j.jvir.2017.02.033. Epub 2017 Mar 30. PMID 28365171
- [Background] Okuno Y, Korchi AM, Shinjo T, Kato S. Transcatheter arterial embolization as a treatment for medial knee pain in patients with mild to moderate osteoarthritis. Cardiovasc Intervent Radiol. 2015 Apr;38(2):336-43. doi: 10.1007/s00270-014-0944-8. Epub 2014 Jul 4. PMID 24993956
- [Background] Iwamoto W, Okuno Y, Matsumura N, Kaneko T, Ikegami H. Transcatheter arterial embolization of abnormal vessels as a treatment for lateral epicondylitis refractory to conservative treatment: a pilot study with a 2-year follow-up. J Shoulder Elbow Surg. 2017 Aug;26(8):1335-1341. doi: 10.1016/j.jse.2017.03.026. PMID 28734535
- [Background] Okuno Y, Iwamoto W, Matsumura N, Oguro S, Yasumoto T, Kaneko T, Ikegami H. Clinical Outcomes of Transcatheter Arterial Embolization for Adhesive Capsulitis Resistant to Conservative Treatment. J Vasc Interv Radiol. 2017 Feb;28(2):161-167.e1. doi: 10.1016/j.jvir.2016.09.028. Epub 2016 Dec 19. PMID 28007330
- [Background] Okuno Y, Oguro S, Iwamoto W, Miyamoto T, Ikegami H, Matsumura N. Short-term results of transcatheter arterial embolization for abnormal neovessels in patients with adhesive capsulitis: a pilot study. J Shoulder Elbow Surg. 2014 Sep;23(9):e199-206. doi: 10.1016/j.jse.2013.12.014. Epub 2014 Mar 4. PMID 24618195